CLINICAL TRIAL: NCT00905671
Title: Study of Lipid Core Plaque Shift at Sites of Native Coronary Artery Bifurcation
Brief Title: Intravascular Near Infrared Spectroscopy (NIRS) Bifurcation - Lipid Core Plaque Shift Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Infraredx (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0102
Record Dates: First submitted 2009-05-15; First posted 2009-05-20 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Angina Pectoris; Angina, Unstable; Atherosclerosis; Coronary Artery Disease
Keywords: Lipid Core Plaque; LCP; Bifurcation; Stenosis; Lesion; Angioplasty
MeSH Terms: conditions — Angina Pectoris; Angina, Unstable; Atherosclerosis; Coronary Artery Disease; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP+ Bifurcation Lesion (Experimental): Bifurcating lesions that are positive for lipid core plaque, as detected by LipiScan Coronary Imaging, prior to angioplasty.
  Interventions: Device: LipiScan Coronary Imaging Catheter
- LCP- Bifurcation Lesion (Experimental): Bifurcating lesions that are not positive for lipid core plaque, as detected by LipiScan Coronary Imaging, prior to angioplasty.
  Interventions: Device: LipiScan Coronary Imaging Catheter

INTERVENTIONS:
Device: LipiScan Coronary Imaging Catheter — Intravascular near infrared spectroscopic imaging of the coronary artery with a fiberoptic catheter.

SUMMARY:
This pilot study is going to examine the hypothesis that in coronary arteries, soft lesions that contain lipid cores, but are not calcified or fibrotic and are located in proximity to side branches, are associated with side branch compromise as a result of plaque shift during angioplasty and stenting. Plaque characteristics will be detected by intravascular near infrared spectroscopy (NIRS).

DETAILED DESCRIPTION:
Coronary artery bifurcations (branching areas) are predisposed to atherosclerosis from turbulent flow and increased shear stress. Dilating lesions that involve a branch vessel is associated with the risk of closure of the side branch. Plaque redistribution or 'plaque shift' across the carina of the bifurcation is regarded as the responsible mechanism for the side branch stenosis and occlusion after angioplasty and stenting. Modern techniques of side branch protection require positioning of a second wire into the side branch before starting the treatment of the main branch. Placing an additional wire in the side branch is more laborious and complex than the wiring of the main branch only, is associated with additional use of contrast media and radiation, and may associated with additional risk of complications. Being able to determine which side branches require wiring for protection while treating the main vessel stenosis may make the procedure simpler and safer.

Lipid core plaque (LCP) in the coronary arteries is very common in acute coronary syndrome, but can often be found also in patients with stable angina. Lipid core plaque cannot be detected by angiography or intra-vascular ultrasound. Near infrared spectroscopy (NIRS) has the ability to identify chemicals in mixture. LipiScan, a catheter based NIRS coronary imaging system can detect intra-vascular LCP. This catheter has been shown to be able to identify LCP through blood in a prospective autopsy study, and that the LCP detection algorithm developed and validated on ex vivo data is applicable in vivo. The image generated by this system is called 'chemogram'. The catheter has also been tested successfully in a clinical study in the United States and Canada. Based on these studies the FDA approved the use of the LipiScan coronary imaging system. In CUMC, we have started to use this catheter to identify LCP, and have gained experience with its simple use.

This study is intended as a pilot study to identify angioplasty related redistribution or shift of lipid core plaque (LCP) lesions that are located at sites of artery bifurcation. We hypothesize that during angioplasty and stenting, soft plaque that contains lipid cores may be prone to shift more than (hard) fibrotic or calcified lesions. This pilot study may help to better characterize lesions likely to shift and to provide imaging-based information like NIRS that will improve the interventional treatment of bifurcation lesions.

A total of 20 patients with significant coronary artery disease with a bifurcation lesion suitable for angioplasty and stenting will be studied. The lesions that will be studied contain significant stenosis (≥50% stenosis) located in proximity (less than 2 mm) to a side branch. Prior to angioplasty, the main vessel involved in the bifurcation will be imaged using the LipiScan Coronary Imaging System. Angioplasty and stenting will be performed in the usual conventional way, and then re-imaged with the LipiScan system. Intravascular ultrasound will be done as standard interventional imaging procedure, when directed by the treating interventional cardiologist. Angiographic and Chemographic data will be qualitatively and quantitatively analyzed to assess LCP and plaque shift into the side branch. Subjects that have intravascular ultrasound as part of routine care, will have this data analyzed and compared to the chemogram data.

Improved understanding of how plaques and lipid cores redistribute and under what conditions redistribution occurs could assist interventional cardiologists to better plan and perform complex procedures that involve bifurcation plaques. Improved procedural planning and prediction of shift can reduce instances of difficult side branch rescue and reduce occurrence of peri-procedural events, such as myocardial infarction. This may in turn lead to a reduction in overall complexity of treatment procedures, complication, and procedure recovery times.

The catheter-based interventional treatment of branching points in blocked heart blood vessels is complex and prone to higher rate of complications. This study is intended to better understand why and under what conditions coronary blockages move during balloon angioplasty and stenting. The movement of coronary artery blockages during the standard treatment of coronary disease often leads to blocking of small artery branches near the treatment site. The blocking of these small branches does not occur at all times, but when it does occur it often results in small myocardial infarctions or residual chest pain.

All patients in this study will undergo standard cardiac catheterization and intervention as directed by their treating physician. In this research, the researchers will analyze imaging data that will be collected during the procedure. This includes the angiography (all patients), intravascular ultrasound (in the patients that the operator determines its need for use as part of the procedure), and imaging from the LipiScan catheter (all patients). The LipiScan catheter is approved by the FDA for intravascular detection of fat in the blood vessel, and will be used to detect the fat composition of the blockage. This catheter, detects whether the blockage is composed of fat and is soft, or is fibrous and hard. In this study we are going to try to identify the type of blockages that are associated with branching points, and to learn whether soft and fat containing blockages are associated with shifting or movement of the blockage material into the side branch. The information learned from this study may help interventional cardiologists in the future to better plan their interventional techniques and strategy and to perform safer and more successful procedures.

Coronary artery bifurcations (branching areas) are predisposed to atherosclerosis from turbulent flow and increased shear stress. Lesions situated at a bifurcation segment account for up to 16% of the interventional procedures (1). Stenoses at a bifurcation remains one of the most technically challenging lesion subsets to treat by coronary angioplasty and stenting (2- 5). Dilating lesions that involve a branch vessel is associated with the risk of stenosis or complete closure of the side branch. In the past, bifurcation lesions were considered a contraindication to PTCA due to the significantly increased risk of side-branch occlusion. In various series, the rates of side branch stenosis or occlusion post angioplasty and stenting is in the range of 9-67% (6-11) of threatened side branches. Salvage of an occluded side-branch may be difficult, and unsuccessful in around 50% of rescues, especially when the ostium of the side branch contains stenosis prior to occlusion (12, 13). In other cases, the side branch is not occluded, but may be severely narrowed, mainly because of plaque shift. Over the years, with the improved experience, techniques, and technology, it is common practice now to treat bifurcation lesions percutaneously, with high success and acceptable complication rates. Nevertheless bifurcation lesion pose higher technical demand and more use of interventional devices.

Using IVUS imaging, plaque redistribution was described during stenting (14, 15). Plaque redistribution or 'plaque shift' across the carina of the bifurcation is regarded as the responsible mechanism that compromises the side branch lumen. Other predictors of side branch occlusion include significant branch-ostial stenosis, main vessel dissection, and acute coronary syndrome including acute MI (16). The later are important situations in which there may be a combination of thrombus on top of a lipid containing plaque.

Modern techniques of side branch protection entails positioning of a second wire into the side branch before starting the treatment of the main branch (1,16, 17). The decision to protect the side branch depends on the estimated risk of closure while treating the main branch. Unfortunately, it is impossible to predict whether or not a specific side branch will be compromised. Advancing an additional wire in the side branch is more laborious and complex than the wiring of the main branch, mandating the use of larger caliber guiding catheters, prolongs the overall procedure time, associated with larger volume of contrast media and x-ray radiation, and may be associated with increased risk of complications like coronary dissection, perforation, bleeding and contrast induced nephropathy (1). The ability to identify which side branches need to be wired and protected while working on the main vessel will make the procedure simpler and safer.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >=40yrs
* Subject must provide written informed consent.
* Subject must be diagnosed with stable or unstable angina pectoris, or documented silent ischemia
* Subject must be scheduled for elective or non-emergent percutaneous coronary intervention
* Angiographic evidence of a bifurcation lesion with the following characteristics:

  * Native coronary artery
  * De novo coronary stenosis at the bifurcation site
  * Bifurcation Medina class 1,1,0 or 1,0,0 or 0,1,0
  * Main vessel stenosis >50%, with the stenotic lesion in close proximity (≤2mm) to the side branch ostium, by visual estimate.
  * Side branch diameter ≥ 2.0mm by visual estimate.
  * Side branch without significant stenosis (<30% stenosis)
  * LipiScan catheter optical tip must cross lesion without the need for pre-dilatation

Exclusion Criteria:

* Subject is pregnant or nursing
* Renal insufficiency (Creatinine >2.0mg/dL)
* Left ventricular ejection fraction <25% by visual estimate.
* Known allergy to contrast media that cannot be medically managed.
* Acute ST segment elevation myocardial infarction (STEMI) that has not been stabilized.
* Any condition or symptom that in the investigator's opinion may adversely alter the risk profile of this study for the subject.
* Target lesion is dilated prior to first LipiScan imaging.
* Subject experiences procedural complication that precludes clear post angioplasty imaging of the target lesion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Angiographic evidence of plaque shift. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Giora Weisz, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Reimers B, Colombo A, Tobis J. Bifurcation Lesions. In: Colombo A, Tobis J, eds. Techniques in Coronary Artery Stenting. London 2000, pp 171-204.
- [Background] Louvard Y, Lefevre T, Morice MC. Percutaneous coronary intervention for bifurcation coronary disease. Heart. 2004 Jun;90(6):713-22. doi: 10.1136/hrt.2002.007682. No abstract available. PMID 15145893
- [Background] Colombo A, Moses JW, Morice MC, Ludwig J, Holmes DR Jr, Spanos V, Louvard Y, Desmedt B, Di Mario C, Leon MB. Randomized study to evaluate sirolimus-eluting stents implanted at coronary bifurcation lesions. Circulation. 2004 Mar 16;109(10):1244-9. doi: 10.1161/01.CIR.0000118474.71662.E3. Epub 2004 Feb 23. PMID 14981005
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Louvard Y, Lefevre T. Bifurcation lesion stenting. In Colombo A, Stankovic G, eds. Problem oriented approaches in interventional cardiology. Informa Healthcare 2007.
- [Background] Fischman DL, Savage MP, Leon MB, Schatz RA, Ellis S, Cleman MW, Hirshfeld JW, Teirstein P, Bailey S, Walker CM, et al. Fate of lesion-related side branches after coronary artery stenting. J Am Coll Cardiol. 1993 Nov 15;22(6):1641-6. doi: 10.1016/0735-1097(93)90589-s. PMID 8227832
- [Background] Mazur W, Grinstead WC, Hakim AH, Dabaghi SF, Abukhalil JM, Ali NM, Joseph J, French BA, Raizner AE. Fate of side branches after intracoronary implantation of the Gianturco-Roubin flex-stent for acute or threatened closure after percutaneous transluminal coronary angioplasty. Am J Cardiol. 1994 Dec 15;74(12):1207-10. doi: 10.1016/0002-9149(94)90549-5. PMID 7977091
- [Background] Pan M, Medina A, Suarez de Lezo J, Romero M, Melian F, Pavlovic D, Hernandez E, Segura J, Marrero J, Torres F, et al. Follow-up patency of side branches covered by intracoronary Palmaz-Schatz stent. Am Heart J. 1995 Mar;129(3):436-40. doi: 10.1016/0002-8703(95)90264-3. PMID 7872167
- [Background] Aliabadi D, Tilli FV, Bowers TR, Benzuly KH, Safian RD, Goldstein JA, Grines CL, O'Neill WW. Incidence and angiographic predictors of side branch occlusion following high-pressure intracoronary stenting. Am J Cardiol. 1997 Oct 15;80(8):994-7. doi: 10.1016/s0002-9149(97)00591-2. PMID 9352966
- [Background] Bhargava B, Waksman R, Lansky AJ, Kornowski R, Mehran R, Leon MB. Clinical outcomes of compromised side branch (stent jail) after coronary stenting with the NIR stent. Catheter Cardiovasc Interv. 2001 Nov;54(3):295-300. doi: 10.1002/ccd.1287. PMID 11747152
- [Background] Almeda FQ, Nathan S, Calvin JE, Parrillo JE, Klein LW. Frequency of abrupt vessel closure and side branch occlusion after percutaneous coronary intervention in a 6.5-year period (1994 to 2000) at a single medical center. Am J Cardiol. 2002 May 15;89(10):1151-5. doi: 10.1016/s0002-9149(02)02295-6. PMID 12008166
- [Background] Ciampricotti R, el Gamal M, van Gelder B, Bonnier J, Taverne R. Coronary angioplasty of bifurcational lesions without protection of large side branches. Cathet Cardiovasc Diagn. 1992 Nov;27(3):191-6. doi: 10.1002/ccd.1810270307. PMID 1423574
- [Background] Weinstein JS, Baim DS, Sipperly ME, McCabe CH, Lorell BH. Salvage of branch vessels during bifurcation lesion angioplasty: acute and long-term follow-up. Cathet Cardiovasc Diagn. 1991 Jan;22(1):1-6. doi: 10.1002/ccd.1810220102. PMID 1995167
- [Background] Ahmed JM, Mintz GS, Weissman NJ, Lansky AJ, Pichard AD, Satler LF, Kent KM. Mechanism of lumen enlargement during intracoronary stent implantation: an intravascular ultrasound study. Circulation. 2000 Jul 4;102(1):7-10. doi: 10.1161/01.cir.102.1.7. PMID 10880407
- [Background] Maehara A, Takagi A, Okura H, Hassan AH, Bonneau HN, Honda Y, Yock PG, Fitzgerald PJ. Longitudinal plaque redistribution during stent expansion. Am J Cardiol. 2000 Nov 15;86(10):1069-72. doi: 10.1016/s0002-9149(00)01161-9. PMID 11074201
- [Background] Safian RD, Freed MS, Grines C, Freed M. ed., The Manual of Interventional Cardiology. pp 221-236.
- [Background] Louvard Y, Lefevre T, Cherukupalli R. Favorable Effect of the Jailed Wire Technique When Stenting Bifurcation Lesions. Am J Cardiol 2003:6 (abstr, suppl).